CLINICAL TRIAL: NCT03883451
Title: Evaluation of Helmet Technology and Head Impact Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-2799
Record Dates: First submitted 2018-12-27; First posted 2019-03-21 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: MTBI - Mild Traumatic Brain Injury; Concussion, Mild
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: single group of football athletes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Helmet type (Experimental): football player helmet model
  Interventions: Other: Helmet Model

INTERVENTIONS:
Other: Helmet Model — helmet model worn by football players

SUMMARY:
The purpose of the study is to monitor longitudinal changes in brain structure and function between the preseason and postseason, in a population of football playing athletes grouped by helmet make and model. Secondly, the purpose is to determine the protection of the helmet make and model relative to amount and magnitude of sustained head impacts.

DETAILED DESCRIPTION:
Sports-related traumatic brain injury (sTBI) is common in competitive sports and recreational activities, with 1.6 to 3.8 million reported annually in the U.S. Children, adolescents and young adults are at the highest risk for sustaining mild TBI. There is scarce high-level prospective, objective evidence indicating that any recent helmet design can prevent sTBI. While helmets were developed for, and are effective in, preventing skull fractures and intracranial hematomas, it is unclear if they afford protection against forces inside the cranium.

This study will investigate the relationship between potential changes in brain structure and function pre and post season compared to helmet make and model and head impact exposure in high school and college athletes playing a collision sport such as football. The use of helmets/headgear during such a high-risk sport will allow for collision measurement devices to be affixed to the athlete under the helmet and will not affect play or fit of equipment. By the nature of the sport selected, it is likely this study will primarily include males, however if any female meets inclusion criteria on the team selected, the participant will be included in this investigation. All participants will be outfitted with an accelerometer which will measure the magnitude of every impact to the head sustained by the athlete. Effectiveness of the helmet model will be determined via differences in longitudinal brain imaging and functional testing following competitive football participation. A subset of athletes who report a diagnosed concussion will also receive additional brain neuroanatomical and neurophysiological testing within a week following the diagnosed concussive event. The investigators will also enroll a group of athletes involved in a non-contact sport (such as cross country) to act as controls.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer
* Able to provide written consent
* Must be 13 years or older and a participant on a high school or collegiate team

Exclusion Criteria:

* Unable to provide written consent
* Not medically cleared to participate on a high school or collegiate team

Ages: 13 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Change in brain DTI | 6 months
  change in DTI scan of the brain from pre to post season scans targeting specific regions of interest

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Cincinnati Childrend Hospital
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No